CLINICAL TRIAL: NCT05713149
Title: Treatment of Osteomyelitis-associated Pressure Ulcers by Surgical Flaps and Anti-bacterial Agents in Patients Patients With Neuromotor Disability : a Prospective Cohort Study
Brief Title: Treatment of Osteomyelitis-associated Pressure Ulcers by Surgical Flaps and Anti-bacterial Agents
Status: Recruiting | Type: Observational
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-001
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Disability or Chronic Disease Leading to Disablement; Pressure Ulcer; Osteomyelitis
Keywords: Disability, Pressure Ulcer, Osteomyelitis, Surgical Flaps, Anti-bacterial agents, Posture
MeSH Terms: conditions — Pressure Ulcer; Osteomyelitis | interventions — Surgical Flaps; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with osteomyelitis-associated pressure ulcers: Subjects with neuromotor disability and admitted for the treatment of osteomyelitis-associated pressure ulcers
  Interventions: Other: Surgical flap and anti-bacterial agents

INTERVENTIONS:
Other: Surgical flap and anti-bacterial agents — Surgical flap and anti-bacterial agents

SUMMARY:
People with neuromotor disability (i.e. following an inborn or acquired spinal cord, cerebral or peripheral neurological lesion) are at high risk of osteomyelitis-associated pressure ulcers.

The management of osteomyelitis-associated pressure ulcers is controversial. In our center, patients benefit from a one stage surgical management with bone shaving and flap covering osteitis of pressure ulcer to perform wound closing. Surgery is followed by an antibiotic treatment, secondarily adapted to intraoperative samples.

The aim of this study is to describe the cohort and to identify factors associated with failure (or success) in this frail population.

DETAILED DESCRIPTION:
This is a prospective, monocentric, cohort study of neurological disabled inpatients subjects treated in the perioperative disability unit (UPOH) of our university hospital for osteomyelitis-associated pressure ulcer by surgical flaps and anti bacterial agents.

All eligible inpatient subjects with neuromotor disability and admitted for the treatment of osteomyelitis-associated pressure ulcers by surgical flaps will be consecutively included.

Patients are followed up in consultation at 30 or 45 days after surgery, and in consultation or teleconsultation at 12 months after surgery.

Data will be collected from the patients' medical records, in particular data related to their clinical, radiological, biological, and physiological examinations. Data related to sitting, nutrition, spasticity, bladder and bowel disorders, bacteriological sampling and antibiotic treatments will be collected.

This is a routine care study; no procedures are added for research purposes. It is an ancillary study to the NO-AGING study.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old ;
* Treated in the Perioperative Disability Unit (UPOH) of the Physical Medicine and Rehabilitation Department of our university hospital;
* Admitted for the treatment of an osteomyelitis-associated pressure ulcer by surgical flap;
* Having a neuromotor disability;
* No opposition to be enrolled in the study from the patient, or from a legally authorized close relative if the patient's state of health does not allow it;
* Affiliation to a social security scheme.

Exclusion Criteria:

* Under court protection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with neuromotor disability and admitted for the treatment of osteomyelitis-associated pressure ulcers by surgical flaps and antibacterial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-19 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Success at 12 months after surgery | 12 months after surgery
  Success is defined as the absence of surgical revision, the absence of additional antibiotic therapy, and the absence of local care at the surgical site.

SECONDARY OUTCOMES:
Success at 30-45 days after surgery | 30-45 days after surgery (depening on the surgical technique)
  Success is defined as the absence of surgical revision, the absence of additional antibiotic therapy, and the absence of inflammatory signs or pus leakage or deep disunion of more than 2 cm.
Description of the patients' bacteriological tests | Through hospital admission, up to 7 days after surgery
  Intraoperative samples and drain samples.
Death | 12 months after surgery
  Obtained from the INSEE database.

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD-PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garches, France

IPD SHARING:
Plan to Share IPD: No